CLINICAL TRIAL: NCT02187419
Title: Hypnosis to Improve Sleep in Menopause: Determination of Optimal Dose and Method
Brief Title: Hypnosis to Improve Sleep In Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Responsible Party: Principal Investigator, Gary R. Elkins, PhD, Baylor University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R34AT008246-01 (NIH)
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Sleep
Keywords: Sleep; Menopause; Hypnosis; Relaxation; Hypnotic Relaxation Therapy; Hot Flash
MeSH Terms: conditions — Hot Flashes | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 5 Therapist-Delivered Hypnosis Session (Active Comparator): Participants will complete five therapist-delivered hypnosis relaxation sessions with a hypnosis research therapist, and receive five audio (CD or MP3) recordings of hypnotic inductions and instructed in daily home practice.
  Interventions: Other: Hypnosis
- 3 Therapist-Delivered Hypnosis Session (Active Comparator): Participants will complete three therapist-delivered hypnosis relaxation sessions with a hypnosis research therapist, and receive five audio (CD or MP3) recordings of hypnotic inductions and instructed in daily home practice.
  Interventions: Other: Hypnosis
- 5 Phone Calls; Hypnosis Recordings Only (Active Comparator): Participants will complete five phone calls with a hypnosis research therapist, and receive five audio (CD or MP3) recordings of hypnotic inductions and instructed in daily home practice.
  Interventions: Other: Hypnosis
- 3 Phone Calls; Hypnosis Recordings Only (Active Comparator): Participants will complete three phone calls with a hypnosis research therapist, and receive five audio (CD or MP3) recordings of hypnotic inductions and instructed in daily home practice.
  Interventions: Other: Hypnosis

INTERVENTIONS:
Other: Hypnosis — Hypnosis is a promising, but under-studied non-pharmacological treatment option for poor sleep during the menopausal transition. Hypnosis is a mind-body therapy that may be defined as a deeply relaxed state involving mental imagery and suggestion. The hypnotic state has been described variously as being an altered state of consciousness, focused attention, imaginative involvement, and role assumption.
  However, it is generally agreed that hypnosis is a "state or condition, which occurs when appropriate suggestions elicit distortions of perception, memory, or mood". Research has shown that most people are hypnotizable. Hypnosis intervention for managing chronic symptoms usually involves a hypnotic induction, instruction in self-hypnosis and practice using audio recordings.
  Other Names: Hypnotic Relaxation Therapy

SUMMARY:
The purpose of this study is to determine feasibility and adherence to a hypnosis program to improve sleep. It is theorized (based on prior experience and pilot data) that one or more hypnosis program(s) will be feasible and will exhibit acceptable adherence. The programs will assess to determine optimal dose (3 vs 5 sessions) and method (audio-recorded vs therapist delivered).

DETAILED DESCRIPTION:
It is conceptually theorized that one or more hypnosis program(s) [dose and delivery] will be feasible and will exhibit acceptable adherence to daily hypnosis practice to improve sleep. The optimal dose (3 vs. 5 sessions) and delivery method (audio recorded vs. therapist delivered) are as yet unknown. It is hypothesized that a hypnosis program will indicate an effect on objectively measured sleep duration. It is expected that one or more hypnosis interventions will have effects on both the primary outcome (objectively measured sleep duration) and secondary outcomes (sleep quality, insomnia symptom severity, daytime sleepiness, menopausal symptoms, pain, and bothersomeness).

This study will provide estimated effect sizes for the primary and secondary outcomes for later studies. In addition, it is possible that there are potential covariates such as age, race, menopausal stage, sleep environment, and/or socioeconomic status that require consideration. These will be explored (Aim 4) to guide the future, larger study.

Stratified randomization will be utilized, with one variable present in the randomization: the presence/absence of hot flash . "Presence" of hot flash is determined by criteria used in a prior study (i.e., 7 hot flashes per day, or 50 hot flashes per week) during the screening or baseline week. If the criteria is not met that indicates presence of hot flashes and reported during those two weeks, then the woman will be determined as not having hot flashes.

Objectives

* Aim 1: Determine the feasibility of and adherence to the four hypnosis programs. Feasibility will be determined by (1) a dropout rate of less than 25%, (2) participants' rating of the program (from poor to excellent; with rating of good or better defined as feasible), (3) participants' rating of treatment satisfaction (from completely satisfied to completely dissatisfied) and (4) few adverse events (<5%). Adherence will be determined through daily at-home practice forms. An adherence threshold of 75% will be utilized as this level of adherence is likely to be needed for an optimal hypnosis program for sleep.
* Aim 2: Determine initial effect sizes for the primary outcome of objectively measured sleep duration, including the percent of women who achieve a clinically meaningful improvement. Wrist actigraphy recordings supplemented by sleep diaries will be used to measure sleep duration. Clinically meaningful improvement is defined as the percentage of women who move from poor to average sleep duration (e.g., from < 6.5 hours per night to > 6.5 hours but <9.0 per night).
* Aim 3: Determine initial effect sizes for secondary outcomes of sleep quality, insomnia symptom severity, daytime sleepiness, menopausal symptoms, and pain.
* Aim 4: Examine trends in potential covariates including endogenous factors (e.g., age, race/ethnicity, menopausal status) and exogenous factors (e.g., sleep environment, socioeconomic status).

Study Design

This study is designed as a 4-arm comparison, with participants randomized to the following arms:

1. Standard audio recordings for home practice, with 5 in-person therapist delivered hypnotic inductions
2. Standard audio recordings for home practice, with 3 in-person therapist delivered hypnotic inductions
3. Standard audio recordings only, with 5 telephone contacts to encourage home practice
4. Standard audio recordings only, with 3 telephone contacts to encourage home practice

ELIGIBILITY:
Inclusion criteria are:

* Females, aged 40-65. (This proposed range is based on the Menopause Strategies: Finding Lasting Answers for Symptoms and Health (MsFLASH) criteria to identify symptomatic women in the menopausal transition and to allow for comparison to other studies of this target population)
* Self-reported sleep duration of ≤6 hours per day/night for 5 or more nights per week as determined by a 7-day sleep diary during screening and baseline weeks
* Post-menopausal or in the late perimenopausal transition, defined as ≥ 2 missed menstrual cycles with an interval of amenorrhea ≥ 60 days in the past 12 months
* In general good health as determined by medical history and physical measures
* Non-depressed as determined by Patient Health Questionnaire (PHQ-8) scores ≤ 9
* Signed informed consent

Exclusion criteria are:

* Use of hormone therapy or hormonal contraceptives during the 2 months before enrollment and for the duration of the study
* Self-report of sleep apnea and/or restless leg syndrome
* Use of any prescription or over-the-counter therapy for sleep (i.e. Melatonin, valerian, other "natural" sleep aids, and commonly used over-the-counter (OTC) medications [e.g. acetaminophen + diphenhydramine or equivalent]) [NOTE: Medications not intended for sleep but that have a known impact on sleep will be allowed (i.e. serotonin-norepinephrine reuptake inhibitors-SNRIs, selective serotonin re-uptake inhibitors-SSRIs)]
* Severe or unstable medical or psychiatric illness
* Current use of hypnosis for any condition
* Inability to speak or understand English [NOTE: Providing hypnosis is highly dependent on the use of language. While it would be possible to recruit a Spanish speaking hypnotherapist, none of the investigators speak Spanish and this would make it extremely difficult (if not unethical) to provide supervision to a Spanish speaking hypnotherapist. Because of this we have elected to restrict participants to those that are English speaking]

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-02-24 (Actual)

PRIMARY OUTCOMES:
Objective sleep duration | Eight weeks
  Wrist actigraphy: Wrist actigraphy is a widely used and well-validated, objective measure of sleep duration. Participants will be asked to wear an Actiwatch 2; Phillips Respironics, which resembles a wrist watch, on their non-dominant wrist. A motion detection device located within the actigraph records movement. After data is collected it will be analyzed using a software program which uses a series of logarithms to measure various factors associated with sleep quality, such as total sleep duration, sleep efficiency, sleep onset latency, and the number of times participants woke during the night. Wrist actigraphy has been used to reliably differentiate the sleeping patterns of men and women. For the present study, participants will be asked to wear the actigraph from baseline assessment throughout the study through week eight.
  Participants will also complete a Daily Sleep Diary that will be used to help interpret wrist actigraphy data.

SECONDARY OUTCOMES:
PHQ-8 | Screening
  The PHQ-8, an 8-item depression scale, is an established measure of depression and has been validated in large clinical studies as well as among primary care and obstetrics-gynecology outpatients. It is an excellent severity, diagnostic, and monitoring measure, and will be used to screen for depression, using the cutpoint of ≥ 9 to define current depression for this study.
Pittsburgh Sleep Quality Index (PSQI) | Baseline, Week 4, Week 6, Week 8
  The PSQI is a 19-item self-report inventory designed to measure sleep quality. The 19 items are grouped into 7 subscales: 1) sleep quality, 2) sleep efficiency, 3) daytime dysfunction, 4) sleep latency, 5) sleep disturbances, 6) sleep duration, and 7) use of sleep medication. These seven subscales are scored on a scale of 0-3 with higher scores indicating greater sleep pathology. Global scores above 4 are normally considered indicative of poor sleep quality. Previous studies indicate that PSQI total scores are significantly correlated with measures of sleep onset latency, amount of time spent awake after initial sleep onset, and total sleep time as assessed by sleep diary and wrist actigraphy, and alphas for the PSQI range from .70 to .80.
Insomnia Severity Index (ISI) | Baseline, Week 4, Week 6, Week 8
  The ISI consists of seven items that measure the severity of sleep onset, sleep maintenance, and early morning awakening problems, as well as the participant's satisfaction with her current sleep pattern, the extent to which lack of sleep interferes with daily functioning, how noticeable this impairment is to other people, and the extent to which the participant is worried or distressed about their lack of sleep. Items are scored on a scale from 0-4 with total score of 15 or higher indicating the presence of clinical insomnia. Past research indicates that internal reliability estimates for the ISI range from .74 to .78, and correlations between individual items from the ISI and diary reports for sleep onset latency, time awake after initial sleep onset, and time awake before rising from bed are all significant at the p < .001 level.
Epworth Sleepiness Scale (ESS) | Baseline, Week 4, Week 6, Week 8
  The ESS is an 8-item self-report measure that asks participants to indicate how likely they are to fall asleep while engaging in eight different everyday activities (e.g. watching television, sitting in traffic). Items are scored on a scale from 0-3 with higher scores indicating a greater probability of falling asleep. Previous research indicates that the ESS has a Cronbach's alpha of .88 and also that ESS scores correlate significantly with polysomnography ratings of sleep-latency.
Menopausal Rating Scale (MRS) | Baseline, Week 4, Week 6, Week 8
  The MRS is an 11-item self-report measure that asks participants to rate the severity of 11 different menopausal symptoms (including hot flashes) on a scale from 0-4, with higher scores indicating greater symptom distress. The 11 items on the MRS are divided into three subscales; psychological, somato-vegetative, and urogenital. Previous research indicates that the MRS has a Cronbach's alpha of .88 when used with American women and that MRS scores are highly correlated with both Kupperman ratings and Short-Form-36 subscale scores.
Pain Visual Analog Scale (VAS) | Baseline, Week 4, Week 6, Week 8
  Participants will be asked to rate their pain on a 10-cm VAS during baseline assessment and at weeks four, six, and eight of the study. Participants will be asked to place an "X" along the 10-cm line to indicate the severity of their pain over the past week, with the lower (left) end of the scale being anchored by the phrase "no pain" and the upper (right) end of the scale being anchored by the phrase "the most intense pain possible". Previous work indicates that visual analog scales provide researchers with a highly reliable and valid method of assessing pain in adult women.
Bothersomeness Numeric Rating Scale (NRS) | Baseline, Week 4, Week 6, Week 8
  Participants will be asked to assess the degree to which their sleep problems are bothersome using a 0 (not at all) to 10 (extremely)-point NRS. The NRS has good sensitivity and provides data that can be statistically analyzed for research purposes.
Demographic Questionnaire | Baseline
  Demographic data will be collected as potential covariates including age, marital status, socioeconomic status, eligibility for the study, menopausal status, presence of hot flashes or not, and other demographic information
Sleep environment | Baseline, Week 4, Week 6, Week 8
  Data on sleep environment will be collected as a potential covariate on the Sleep Environment Questionnaire. This information will be collected at baseline as well as at weeks four, six, and eight; which will allow us to examine any trends in changes in sleep environment.

CONTACTS AND LOCATIONS:
Overall Officials: Gary R Elkins, PhD, Principal Investigator — Baylor University
Locations (1):
- Mind-Body Medicine Research Lab-Baylor University, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elkins GR, Fisher WI, Johnson AK, Carpenter JS, Keith TZ. Clinical hypnosis in the treatment of postmenopausal hot flashes: a randomized controlled trial. Menopause. 2013 Mar;20(3):291-8. doi: 10.1097/gme.0b013e31826ce3ed. PMID 23435026
- [Background] Elkins G. Hypnotic Relaxation Therapy: Principles and Applications. New York, NY: Springer Publishing Company; 2013.
- See also: Gary Elkins, Baylor University, Department of Psychology & Neuroscience, School of Arts & Sciences — http://www.baylor.edu/psychologyneuroscience/index.php?id=69753